CLINICAL TRIAL: NCT01571323
Title: Combined Use of Oxytocin and Misoprostol Versus Oxytocin Infusion and Misoprostol Alone to Reduce Blood Loss at Cesarean Section
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, assistant professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12612000095864
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Post Partum Haemorrhage
Keywords: post partum haemorrhage at cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin
- Oxytocin and Misoprostol (Active Comparator)
  Interventions: Drug: Oxytocin and Misoprostol

INTERVENTIONS:
Drug: Misoprostol — The misoprostol group (groupM) received 400 µg sublingually and infusion of lactated Ringer ( which one ampoule placebo dissolved it)
  Arms: Misoprostol
Drug: Oxytocin — The oxytocin group(group O) received intravenous infusion of 20 units of oxytocin soon after delivery of the neonate and one tablet of placebo sublingually. (20 IU syntocinon dissolved in 1liter of lactated Ringer's solution) at the rate of 1000 ml over a 1h period, immediately after delivery of the neonate
  Arms: Oxytocin
Drug: Oxytocin and Misoprostol — The combined misoprostol-oxytocin group(group MO) received 200 µg and 5 iu oxytocin bolus intravenously immediately after delivery of the neonate .
  Arms: Oxytocin and Misoprostol

SUMMARY:
The purpose of this study is to demonstrate that the combined used of low dose of oxytocin and misoprostol prevent from post partum haemorrhage better than oxytocin or misoprostol alone at cesarean sectionOne hundred fifty women with singleton term pregnancy undergoing elective or emergency lower segment cesarean section under spinal anesthesia were included in this study. The patients were randomly allocated to one of three groups of 50 each. The oxytocin group(group O) received intravenous infusion of 20 units of oxytocin soon after delivery of the neonate and one tablet of placebo sublingually. (20 IU syntocinon dissolved in 1liter of lactated Ringer's solution) at the rate of 1000 ml over a 1h period, immediately after delivery of the neonate ,The misoprostol group (groupM) received 400 µg sublingually and infusion of lactated Ringer ( which one ampoule placebo dissolved it) and the combined misoprostol-oxytocin group(group MO) received 200 µg and 5 iu oxytocin bolus intravenously immediately after delivery of the neonate . The main outcome measures were blood loss at cesarean section, change in hemoglobin levels, need for additional oxytocics and drug related side effects.The volume of blood in the suction bottle was measured, blood soaked sponges and added to volume from suction bottle. Hemoglobin values were determined both before surgery and 24 h following surgery. Hemodynamic variables were recorded every 5 minutes during surgery .The need for additional oxytocic therapy, operating time, infusion volume given intraoperatively, need for blood transfusion, side effects of study drug and any significant puerperal morbidity were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term (37-40 wks) gestation scheduled for either elective or emergency lower segment cesarean section

Exclusion Criteria:

* women with any risk factor
* associated with an increased risk of postpartum
* hemorrhage were excluded i.e. anemia (Hb8 g%), multiple gestation, antepartum hemorrhage,poly-hydramnios, two or more previous cesarean sections and/or a history of previous rupture uterus.
* current or previous history of significant disease including heart disease, liver, renal disorders or known coagulopathy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
changes in hemoglobin levels after delivery | Hemoglobin values will be determined both before surgery and 24 h following surgery

SECONDARY OUTCOMES:
Hemodynamic variables | every 5 minutes during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin Medical University Science, Qazvin, Qazvin Province, Iran